CLINICAL TRIAL: NCT03373838
Title: Opposition to Diagnostic or Therapeutic Procedures by Aged Hospitalized Patient on Geriatrics Department.
Brief Title: Opposition to Diagnostic or Therapeutic Procedures by Aged Hospitalized Patient
Acronym: OPTAH
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Thomas TANNOU, Medical Doctor, Centre Hospitalier Universitaire de Besancon
Other Study IDs: P/2017/349
Record Dates: First submitted 2017-11-22; First posted 2017-12-14 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Aging; Refusal, Treatment; Qualitative Research; Epidemiology
MeSH Terms: conditions — Treatment Refusal | interventions — Censuses

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Census: Epidemiological study. Sociodemographic and medical survey.
  Interventions: Other: Census
- Qualitative interview: Individual qualitative interview.
  Interventions: Other: Census

INTERVENTIONS:
Other: Census — Survey and interview
  Other Names: Qualitative study

SUMMARY:
The main object is to identify and understand why some hospitalized aged patients oppose himself to treatment or diagnosis procedure. This mixed study will used a census in a geriatrics department and a qualitative research.

DETAILED DESCRIPTION:
To complete qualitative study, interview will also be conducted with : patients, general practitioner, relative and home carers. An observation of geriatric multidisciplinary staff will be done for better understanding of complexity.

ELIGIBILITY:
Inclusion Criteria:

* geriatric department inpatient.
* presenting opposition to medical or diagnosis procedure
* covered by French Social Security System
* agreed to participate to the study

Exclusion Criteria:

* They did not express himself an opposition
* They disagree to participated
* For qualitative research only : major neurocognitive disorder (MMSE <10).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized patient presenting opposition to medical or diagnosis procedure define as :
  * Repeated expression (at least 2 times to 2 differents professionnals) without agreed between these 2 oppositions.
  * Concerning : medication, invasive diagnosis procedure or withdrawal of catheter.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
30 individual semi-structured interviews | 1 year
  Qualitative data analysis and theorical saturation

SECONDARY OUTCOMES:
100 demographic survey | 1 year
  Statistical analysis
100 medical survey | 1 year
  Statistical analysis

CONTACTS AND LOCATIONS:
Overall Officials: Regis AUBRY, MD/PhD, Study Chair — CHU DE BESANCON; Thomas TANNOU, MD, Principal Investigator — CHU DE BESANCON
Locations (1):
- Centre Hospitalier Universitaire, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tannou T, Trimaille H, Mathieu-Nicot F, Koeberle S, Aubry R, Godard-Marceau A. Investigation of opposition to diagnostic or therapeutic procedures in older people hospitalized in acute geriatric services: the OPTAH pilot study protocol. Pilot Feasibility Stud. 2020 Dec 14;6(1):194. doi: 10.1186/s40814-020-00742-7. PMID 33308277